CLINICAL TRIAL: NCT00339547
Title: Risk Factors for Uterine Fibroids: A Case Control Study and Follow-up Amendment to Study Disease Progression
Brief Title: Risk Factors for Uterine Fibroids: A Case Control Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999995048; OH95-E-N048
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-07-25 (Actual); Status verified 2019-07-23

CONDITIONS: Uterine Fibroids
Keywords: Leiomyomas; Ultrasound; Hysterectomy; Epidemiology; Hyperinsulinemia
MeSH Terms: conditions — Leiomyoma; Hyperinsulinism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The proposed study is designed to estimate the proportion of 35-49 year-old women in a large urban health plan who have had fibroids. The membership of the health plan is approximately 45% black, so estimates for black and white women can be compared. Risk factors for the condition will be studied, and uterine tissue from women having hysterectomies or myomectomies will be studied to identify genetic, hormonal, and protein mediators of tumor growth.

A randomly selected sample of about 1800 women age 35-49 who are members of the George Washington University Health Plan will be invited to participate. Presence of leiomyomas for premenopausal participants with no prior diagnosis of leiomyoma will be determined by an ultrasound examination. Presence of leiomyomas for premenopausal women who report a prior diagnosis of fibroids will be determined by ultrasound evidence in their medical record when available, and by self-report when not available. History of fibroids in postmenopausal women will be based on pathology records for those with surgical menopause and on radiology records or self-report for the small number of naturally postmenopausal women. Estimates of the proportion who have or have had fibroids will be compared for blacks and whites.

To examine risk factors for leiomyoma we will conduct a case-control analysis. Cases will be those women identified with leiomyoma from the random sample, supplemented by women in the same age range who have hysterectomies or myomectomies during the study period and hose excised uteri show evidence of fibroids on standard pathology examination. Women from the random sample with ultrasound or pathology evidence showing no uterine fibroids will constitute the control group. Controls will be compared to cases grouped by size of largest fibroid and grouped by clinical.

A telephone interview and self-administered questionnaire will provide information on demographic factors, medical history, dietary intake, reproductive history, life style factors, and occupational/environmental exposures. Blood will be collected from premenopausal women to measure lipids, insulin, and potential susceptibility genes. Urine will also be collected from premenopausal women early in their menstrual cycles to measure gonadotropin levels. Blood pressure, heart rate, weight, height, and waist-to-hip ration will be measured. Tissue from surgical specimens will be use by collaborators at NIEHS to measure cell proliferation and apoptosis, genetic factors, estrogen and progesterone receptor levels, protein markers of estrogen action, and growth factors.

DETAILED DESCRIPTION:
Uterine leiomyomas are the leading cause of hysterectomy in the United States, accounting for over 200,000 procedures each year. Leiomyoma is a common condition with many tumors being asymptomatic. It is not known which women who have fibroids will develop clinical symptoms. In 1996-1999 the NIEHS Uterine Fibroid Study enrolled 1245 randomly selected premenopausal women, aged 35 to 49, who had been randomly selected from the membership roles of George Washington University Health Plan, a large prepaid health plan in Washington, D.C. Slightly over half of the participants were African American. Participants were asked about prior diagnoses of uterine leiomyomas, and 87% were examined by abdominal/transvaginal ultrasound to screen for uterine leiomyoma. Sixty-two percent of the 1245 had either had a prior diagnosis of leiomyoma or had sonogram evidence of the condition.

Study Objectives:

1. Monitor fibroid-related symptoms over time (Two follow-ups over a five-year period).
2. Measure the proportion of women who undergo major medical intervention (hysteroscopic resection, uterine artery embolization, laser coagulation, myomectomy, or hysterectomy).
3. Identify risk factors for increased symptom severity.
4. Identify risk factors for treatment intervention.

Methods: Premenopausal participants in the Uterine Fibroid Study (1996-1999) will be recontacted twice during the years 2001 - 2005 to obtain information about leiomyoma-related symptoms and medical or surgical treatments. Data will be collected with a computer-assisted telephone interview. Medical records of ultrasound or MRI examinations and major medical or surgical interventions will be abstracted to verify medical follow-up and treatment.

Significance: The presence of leiomyomas can be identified with ultrasound screening when the condition is asymptomatic. However, no data are available that allow clinicians to predict which women will experience morbidity. This longitudinal study will trace disease progression, and identify factors related to increased symptom severity and medical/surgical treatment. The findings could then be used to develop a systematic scoring system that can be used to identify women at high risk.

ELIGIBILITY:
* INCLUSION CRITERIA:

All premenopausal women who participated in the initial study are eligible for the current follow-up study.

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1529 (Actual)
Dates: Start 1995-11-01; Study Completion 2019-07-23

CONTACTS AND LOCATIONS:
Overall Officials: Donna D Baird, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Lamminen S, Rantala I, Helin H, Rorarius M, Tuimala R. Proliferative activity of human uterine leiomyoma cells as measured by automatic image analysis. Gynecol Obstet Invest. 1992;34(2):111-4. doi: 10.1159/000292738. PMID 1356890
- [Background] Cramer SF, Patel A. The frequency of uterine leiomyomas. Am J Clin Pathol. 1990 Oct;94(4):435-8. doi: 10.1093/ajcp/94.4.435. PMID 2220671
- [Background] Grover SR, Quinn MA. Is there any value in bimanual pelvic examination as a screening test. Med J Aust. 1995 Apr 17;162(8):408-10. PMID 7746172